CLINICAL TRIAL: NCT06858176
Title: Research on the Brain Glymphatic System of Parkinson's Disease Patients Based on DTI Technology
Status: Not yet recruiting | Type: Observational
Sponsor: The First People's Hospital of Yunnan (Other)
Responsible Party: Principal Investigator, Lu Sa, doc, The First People's Hospital of Yunnan
Other Study IDs: KHLL2025-KY049
Record Dates: First submitted 2025-02-27; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Glymphatic System; Parkinson's Disease (PD); DTI

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patients with early Parkinson's disease and late Parkinson's disease and healthy volunteer
  Interventions: Other: No intervention was implemented in this observational study

INTERVENTIONS:
Other: No intervention was implemented in this observational study — No intervention was implemented in this observational study

SUMMARY:
Synopsis：The brain glymphatic system is a newly discovered anatomical system for removing waste products and maintaining homeostasis in the brain, and its damage is closely related to a variety of neurological diseases. The diffusion tensor image-analysis along the perivascular space (DTI-ALPS) technique has the advantage of being non-invasive and has been shown to be useful for assessing brain glymphatic system function. The purpose of this study is to use DTI-ALPS technology to evaluate the functional changes of the brain glymphatic system in patients with primary Parkinson's disease at different stages of the disease .

Impact:DTI-ALPS technology is a potential imaging indicator for early diagnosis and monitoring of Parkinson's disease progression, and has definite value for clinical application.

Purpose :the functional changes of brain glymphatic system in patients with Parkinson's disease at different stages of the disease will be investigated based on DTI-ALPS technology Methods:The clinical data of 100 patients with primary Parkinson's disease will be admitted to the First People's Hospital of Yunnan Province from March 2025 to April 2026 wil be prospectively collected, and they will be divided into two groups: 50 patients with early Parkinson's disease and 50 patients with late Parkinson's disease according to the Hoehn-Yahr Scale , and 50 healthy volunteers (HC) matched with them will be collected. All subjects will be scanned with a 3.0 T MRI system（MAGNETOM Prisma,Siemens Healthcare,Erlangen,Germany）.The scanning sequences included conventional MRI noncontrast and DTI sequences, which acquired images of b=0 s/mm² and b=1000 s/mm²4. FSL and ITK-SANP software will be used to delineate circular ROIs with voxel diameters of 5 mm in the projection fiber and contact fiber regions at the bilateral ventricular body level of the anisotropy score map, and the diffusivity of each fiber on the x, y, and z axes will be measured, and the DTI-ALPS index value will be calculated, and the one-way ANOVA wii be performed by IBM SPSS statistic 25.0 software, and the differences in the mean ALPS values of the left brain, right brain, and both sides of the subjects in the three groups will be compared. The correlation between the index and clinical data such as age, course of disease, Mini-Mental State Examination Score (MMSE), Montreal Cognitive Assessment Scale, Quality of Life Questionnaire for Patients with Parkinson's Disease (PDQ-39), Parkinson's Disease Non-motor Symptom Evaluation Scale (NMSS), Hamilton Depression Rating Scale score(HAMD), and Unified Parkinson's Rating Scale score (URPDS)will be analyzed.

ELIGIBILITY:
Inclusion Criteria:(1) All the selected candidates were diagnosed in accordance with the "Diagnostic Criteria for Parkinson's Disease in China" (2016 edition) formulated by the International Society of Parkinson's Disease and Movement Disorders and the Parkinson's Disease and Movement Disorders Group and Special Committee of China; (2) Able to cooperate with and tolerate cranial magnetic resonance examination; (3) All are effective against dopamine drugs.

- Exclusion Criteria:(1) secondary parkinsonism (such as after encephalitis, long-term use of neuroleptics such as phenothiazines and butyryls and other drugs such as reserpine, history of toxic exposure, history of vascular diseases such as cerebral infarction or hemorrhage in the basal ganglia, history of traumatic brain injury, abnormal thyroid function, etc.); (2) Parkinson's superposition syndrome (such as progressive supranuclear palsy, olivine pontine cerebellar atrophy, corticobasal ganglia degeneration, Lewy body dementia, Shv. Dräger syndrome, etc.); (3) hereditary degenerative parkinsonism; (4) Patients with diabetes mellitus and end-stage renal disease; (5) Those with contraindications to magnetic resonance examination.

-

Ages: 30 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The clinical data of 100 patients with primary Parkinson's disease will be admitted to the First People's Hospital of Yunnan Province from March 2025 to April 2026 were prospectively collected, and they will be divided into two groups: 50 patients with early Parkinson's disease and 50 patients with late Parkinson's disease according to the Hoehn-Yahr Scale , and 50 healthy volunteers (HC) matched with them will be collected.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
DTI-ALPS | After stopping the medication for 12 hours